CLINICAL TRIAL: NCT01552395
Title: A Prospective Safety Study in 24 Months Treatment of Nocturia With Minirin Melt in Clinical Practice in the Czech Republic
Brief Title: A Study of Minirin Melt in 24 Months Treatment in Patients With Nocturia
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000056
Record Dates: First submitted 2012-03-07; First posted 2012-03-13 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A Confirmation of the Safety Profile for Minirin Melt in Clinical Practice

ELIGIBILITY:
Inclusion Criteria:

* nocturia

Exclusion Criteria:

* habitual or psychogenic polydipsia,
* known or suspected cardiac insufficiency
* other conditions requiring treatment with diuretics
* moderate and severe renal insufficiency
* known hyponatremia
* syndrome of inappropriate ADH secretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients Suffering From Nocturia 1x or More Times a Night
Sampling Method: Non-Probability Sample
Enrollment: 4136 (Actual)
Dates: Start 2012-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 24 months

SECONDARY OUTCOMES:
Number of changes in dosage regime | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (68):
- Czechia (68):
  - Nemocnice Rudolfa a Stefanie (there may be other sites in this country), Benešov
  - Soukromá ambulance, Benešov, Benešov
  - Soukromá ambulance Beroun, Beroun
  - Slezská urologie, Bohunín
  - URIONTEGRITAS soukromá ambulance, Brno
  - Uro - clinic, Brno
  - Urocentrum Brno, Brno
  - Úrazová nemocnice Brno, Brno
  - Soukromá ambalance, Citonice
  - Domažlická Nemocnice, Domažlice
  - Městská nemocnice Dvůr Králové nad Labem a.s., Dvůr Králové nad Labem
  - Nemocnice s poliklinkou Havířov, Havířov
  - Nemocnice Havlíčkův Brod, Havlíčkův Brod
  - Gynekologická ambulance Hluk, Hluk
  - Fakultní nemocnice Hradec Králové, Hradec Králové
  - PPCHC Sanus Hradec Králové, Hradec Králové
  - Městská nemocnice Hustopeče, Hustopeče U Brna
  - Urologická ambulance UROLA, Jaroměř
  - Soukromá ambulance, Jilemnice, Jilemnice
  - Oblastní nemocnice Kladno a.s., Kladno
  - Urologie s.r.o., Klatovy
  - Soukromá ambulance Krnov, Krnov
  - Kromerizska nemocnice a.s., Kroměříž
  - Soukromá ambulance, Lanškroun, Lanškroun
  - Soukromá ambulance Mohelnice, Mohelnice
  - Oblastní nemocnice Náchod, Náchod
  - Sourkomá ambulance, Nový Jičín, Nový Jičín
  - Nemocnice Nový Jičín, Nový Jíčín
  - Centrum MEDIOL s.r.o., Olomouc
  - FN Olomouc, Olomouc
  - Městská nemocnice Ostrava, Ostrava
  - Gynekologická ambulance, Ostrava Ploskovice
  - Vítkovická Nemocnice a.s., Ostrava-Vítkovice
  - Nemocnice Pelhřimov, Pelhřimov
  - FN Plzeň, Pilsen
  - Poliklinika Denisovo nábřeží, Pilsen
  - Nemocnice Písek, Písek
  - Urologická ambulance, Prachatice
  - FN Bulovka, Prague
  - Medicon, Prague
  - Nemocnice s poliklinikou Praha Italská, Prague
  - Soukromá ambulance Praha 7, Prague
  - Soukromá ambulance, Praha 5, Prague
  - Urocare, Prague
  - Urologická klinika Praha 1, Prague
  - Urologické oddělení, Prague
  - Urologie Zahradní Město s.r.o., Prague
  - Urosanté s.r.o, Prague
  - VFN, Prague
  - Ústřední vojenská nemocnice, Prague
  - Urologie - NZZ Lékařský dům, Praha 10 - Uhříněves
  - JR Urocentrum Přerov s.r.o., Přerov
  - Soukromá ambulance, Přeštice, Přeštice
  - Urocare s.r.o., Říčany
  - Soukromá ambulance Štemberk, Štemberk
  - Nemocnice Tábor, Tábor
  - Krajská zdravotní - nemocnice Teplice, Teplice
  - Urologická ambulance, Trutnov
  - Nemocnice Třebíč, Třebíč
  - Nemocnice Podlesí a.s., Třinec
  - Městská nemocnice Turnov, Turnov
  - Nemocnice Uherské Hradiště, Uherské Hradiště
  - Masarykova nemocnice v Ústí nad Labem, Ústí nad Labem
  - Nemocnice Valašské Meziříčí, Valašské Meziříčí
  - DUAM s.r.o. Lékařský dům, Zlín
  - Krajská nemocnice T.Bati a.s., Zlín
  - Soukromá ambulance, Zlín, Zlín
  - UROKAN s.r.o., Znojmo